CLINICAL TRIAL: NCT03861507
Title: Needle Localization During Prostate Brachytherapy Using Power Doppler Ultrasound
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Aaron Fenster, Medical Biophysics Professor, Western University, Canada
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 6442
Record Dates: First submitted 2019-02-28; First posted 2019-03-04 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patient (Other): Patient undergoing standard care prostate high dose rate brachytherapy.
  Interventions: Device: Prostate Brachytherapy

INTERVENTIONS:
Device: Prostate Brachytherapy — High dose - rate (HDR) brachytherapy

SUMMARY:
This study involves patients who are scheduled for standard care brachytherapy of focal tumours within the prostate, which is normally performed under standard 2-dimensional (2D) ultrasound guidance. The purpose of this study is the acquire power Doppler ultrasound while using a simple oscillator in physical contact with the end of a brachytherapy needle. The vibrations along the needle should be visible in the power Doppler ultrasound, helping to visualize the needle position within the anatomy.

ELIGIBILITY:
Inclusion Criteria:

* Male, aged 18 years or older
* Willing to provide written consent
* Pathologically confirmed prostate cancer on previous biopsy
* Suitable for and consenting to high-dose-rate brachytherapy for treatment as standard of care.

Exclusion Criteria:

* • Previous radiotherapy to the prostate

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-03-04 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Needle Trajectory | 1 month following data collection
  Intra-operative needle trajectories in B-mode and power Doppler ultrasound

CONTACTS AND LOCATIONS:
Locations (1):
- Victoria Hospital, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided